CLINICAL TRIAL: NCT02917538
Title: A Randomized Trial of Contact Force in Atrial Flutter Ablation
Acronym: CF-CTIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Mikkel Giehm-Reese, MD, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTIA-2016
Record Dates: First submitted 2016-09-21; First posted 2016-09-28 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2019-11

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): In the intervention group: The operator will perform the RFA treatment guided by real-time CF parameters.
  Interventions: Procedure: RFA
- Control group (Active Comparator): In the control group: The Operator will perform the RFA treatment blinded to the real-time CF parameters.
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — Both groups will receive radiofrequency ablation treatment

SUMMARY:
A clinical randomized trial to evaluate if CF guided Radio Frequency Ablation (RFA) to a specific of LSI in atrial flutter i superior to standard RFA.

DETAILED DESCRIPTION:
Atrial flutter (AFL) is a macro-reentry tachycardia in the right atrium [1,2]. AFL is seen in 0,4 -1,2% of ECG´s in the hospital[3]. Prevalence is higher in patients with structural heart disease, as hypertension, coronary heart disease and cardiomyopathy and also in patients with chronic obstructive lung disease. AFL occurs frequently among patients operated for congenital heart disease.

Cavotricuspid isthmus ablation (CTIA) using radiofrequency (RF) energy is a well-established first line therapy of typical AFL.

The most common arrhythmia requiring treatment is atrial fibrillation (AF). When performing catheter ablation for AF, contact force (CF) applied during radiofrequency energy delivery is a powerful predictor of the electrical isolation of the pulmonary veins and of the clinical response. However, prospective data documenting the superiority of ablation guided by the real time CF monitoring over the standard procedure both for AF and for AFL, are missing. In this regard, showing superiority of ablation guided by the real time CF monitoring over the standard procedure in the simple lesion model of CTIA can serve as a proof of concept for more complex lesion sets, as in AF ablation. The Lesion Size Index (LSI) estimates the size of the lesion created by ablation. It takes account for the nonlinear relationship between the size of the lesion and its three main determinants (CF, power and duration [4,5]), and may therefore be an effective mean to precisely dose the amount of the delivered radiofrequency energy. This may prevent both insufficient lesion creation and complications due to excessive energy delivery. The aim of the present study is to evaluate if CF guided ablation targeting a specific value of LSI is superior to standard radiofrequency catheter ablation (RFCA).

Hypothesis:

CF guided ablation targeting a specific value of LSI is superior to standard RFCA with respect to creating lasting ablation lesions in the cavo-tricuspid isthmus region.

Purpose:

The present study is designed to determine if CF guided ablation targeting a specific value of LSI is superior to standard RFCA with respect to creating lasting ablation lesions in the cavo-tricuspid isthmus region.

Inclusion criteria:

Patients with typical AFL undergoing first CTIA are included.

Exclusion criteria:

Congenital heart disease AF is the dominant arrhythmia Prior right atrial atriotomy Significant mitral valve disease New York Heart Association (NYHA) class IV Secondary AFL (e.g. post-surgery, infections, hyperthyroidism) Age < 40 years Patient does not want to participate.

Study size:

156 patients.

Study design:

Randomized controlled double-blinded study

Inclusion and randomization:

Consecutive patients referred to Department of Cardiology, Aarhus University Hospital, Skejby for ablation of AFL will be screened. All pts without documented AF will undergo a 5 day ambulatory ECG before the scheduled ablation procedure.

Pts with AF documented either on a 12-lead ECG or during ambulatory ECG will be informed about pulmonary vein isolation, if suitable and in the case of accept will be referred for such.

Pts without documented AF fulfilling the inclusion criteria and pts who are not candidates for or not wanting Pulmonary Vein Isolation (PVI) will be invited to an interview with the daily contact person. They will here be informed about the study both orally and written. The interview will take place in a room specially selected for this interview to ensure there will be no interruptions. At the end of the interview pts will be asked to sign a written consent form. Subsequently patients are randomized (computer-based) to two Groups:

1. In group 1, the ablation will be guided by real time CF monitoring and LSI, with a target LSI of 7,0 with a target range 6,8-7.2 . The aim will be a stable contact, and CF 10-30 g. Intermittent contact will be avoided.
2. In group 2, the operator is blinded to the real-time CF.

Randomization Study data are recorded in a web-based case record form (CRF) with loggin of all data entries. The CRF is also used for randomization using computerized permuted blocks of different sizes. Randomization is stratified according to gender. An external data manager is responsible for the CRF and has programmed the random-number generator used.

Follow-up

4 weeks after ablation, a 5 day ambulatory ECG will be performed. 3 months after ablation an Electro Physiological study (EP) will be performed along with administration of adenosine to check the completeness of Bidirectional Isthmus Block (BDIB). In case of reconduction BDIB will be completed. Recurrent isthmus conduction will be classified as located in the anterior half of the isthmus, the posterior half of the isthmus or both.

The follow-up will be 12 months. Patients will be seen at the outpatient clinic 12 month after the ablation, where a 12-lead ECG will be performed. Before this 12 months' visit, a 5 day ambulatory ECG will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical Atrial flutter undergoing first time Cavo Tricuspid Isthmus Ablation

Exclusion Criteria:

* Congenital heart disease
* Atrial fibrillation is the dominant arrhythmia
* Prior right atrial atriotomy
* Significant mitral valve disease
* NYHA IV
* Secondary AFL (e.g. post-surgery, infections, hyperthyroidism)
* Age < 40 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of recurrent isthmus conduction | 3 months
  Rate of recurrent isthmus conduction measured at invasive electrophysiological study 3 months after ablation

SECONDARY OUTCOMES:
Rate of recurrent isthmus conduction in the anterior, middle or posterior third of the isthmus. | 3 months
  Measured at invasive electrophysiological study 3 months after ablation
Freedom from recurrence of Atrial flutter | 3 and 12 months
  Documented by either 12 lead ECG or ambulatory ECG
Occurrence of bidirectional isthmus block with the first ablation line. | 1 hour
  Measured at the primary procedure
Rate of permanent reconduction on the table | 10 minutes
  Rate of permanent reconduction on the table spontaneous and with adenosine within a waiting period of 10 minutes.
Rate of transient reconduction on the table with adenosine | 10 minutes
  Transient reconduction detected by administering adenosine
Ablation time needed to achieve bidirectional isthmus block | 1 hour
  Evaluated at the end of the primary procedure
Total ablation time | 1 hour
  Evaluated at the end of the primary procedure
Total procedure time | 1 hour
  Evaluated at the end of the primary procedure
Quality of Life assesing patients symptoms | 12 months
  Quality of Life assessed by Short-Form-36 (SF-36) questionnaire
Contact Force (CF) | 1 hour
  CF values measured in grams in the two groups
Force-time-integral (FTI) | 1 hour
  FTI values measured in gram seconds in the two groups
Lesion-size-index (LSI) | 1 hour
  LSI values measured in the two groups. LSI does not have a unit but is computed using the FTI value and the power (measured in watts) used during ablation.
Reasons for reconduction | 3 months
  Measuring % of poor ablations for patients with reconduction

CONTACTS AND LOCATIONS:
Overall Officials: Jens Cosedis Nielsen, MD, DMsci, Study Chair — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
We are not authorized to share individual participant data